CLINICAL TRIAL: NCT05969197
Title: Comparative Effects of Match Play Exercises and Plyometric Training on Explosive Power, Agility and Functional Performance in Football Players
Brief Title: Effects of Match Play Exercises and Plyometric Training on Explosive Power, Agility and Functional Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: REC/RCR & AHS/23/0409 Laeeq
Record Dates: First submitted 2023-06-06; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Power; Functional Performance
Keywords: exercise; plyometric; agility; power; functional performance
MeSH Terms: conditions — Motor Activity | interventions — Plyometric Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Match Play Training (Experimental): 15 participants will be in Match play training group giving the Match play exercise protocol along with warm-up sessions for 6 weeks, measuring values before giving them protocol and after protocol.
  Interventions: Other: Match Play Training
- Group B - Plyometric Training (Experimental): 15 participants will be in Plyometric training group giving isotonic exercise protocol along with warm-up sessions for 6 weeks, measuring values before giving them protocol and after protocol.
  Interventions: Other: Plyometric Training

INTERVENTIONS:
Other: Match Play Training — 15 participants will be in Match play training group giving the Match play exercise protocol along with warm-up sessions for 6 weeks, measuring values before giving them protocol and after protocol.
  Arms: Group A - Match Play Training
Other: Plyometric Training — 15 participants will be in Plyometric training group giving isotonic exercise protocol along with warm-up sessions for 6 weeks, measuring values before giving them protocol and after protocol.
  Arms: Group B - Plyometric Training

SUMMARY:
Technique is the most important part of football for scoring goal and in defense of the goal lower limbs are the most important part of the player to be focused on as moving with the ball and training method is important in training football players for their matches. Use of training method in football players can either be a match play training or plyometric training. Plyometric training is considered an effective tool for increasing tendon stiffness. Plyometric training produces improvements in jump performance and lower body strength performance. A training program for young football players, using minimum equipment and effort, can result in improved player performance and a reduction in the risk of a possible overuse injury, reflected by an improvement in lower limb range of motion. Match play training patterns are mostly followed by the coaches to enhance the performance and plyometric are used for the efficient training programs.

This study will be a randomized clinical trial conducted at Pakistan sports board in Lahore. The study will be completed within the time duration of Six months. Non probability convenient sampling technique will be used to collect the data. The sample size of 15 participants each group will be taken in this study to find the effects of match play exercise versus plyometric on explosive power, Agility and functional performance in football players. Football players will be divided into 2 groups Group A will be given the match play training and Group B will be given plyometric trainings and at the end of the 6 week the results will be checked on power, agility and fictional performance. Power: (MRC scale) , Agility: Comprehensive Agility Measurement Tool (CAMT), Functional Performance: The Functional Movement Scale (FMS) tools will be used to measure the difference between the training pattern of 6 weeks which is more effective for the football players. The data will be collected using the SPSS 24. In descriptive statistics Frequency tables, pie charts, bar charts will be used to show summary of group measurements measured over time... The objective of this study is to Determine Comparative Effects of Match play training and plyometric training on Explosive power, Agility and Functional performance in football players.

DETAILED DESCRIPTION:
To Compare the Effects Of Match Play Exercises And Plyometric Training On Explosive Power, Agility And Functional Performance In Football Players Randomized clinical Trials will be used. Non-probability convenient sampling technique will be used Data will be collected from Pakistan Sports Board, Lahore

DATA COLLECTION TOOL

1. POWER Vertical Jump Tests
2. AGILITY Illinois Agility Test
3. The Functional Movement Scale (FMS)

ELIGIBILITY:
Inclusion Criteria:

* • Only Male

  * Ages 15-28(10)
  * Forward , Mid fielders and Defenders (11)
  * Both Right and Left Side players are included

Exclusion Criteria:

* • Lower Extremity Injuries (12)

  * Lower Extremity Deformities
  * History of pain within the previous month prior to testing;
  * Not regular training during the month prior to testing;
  * Musculoskeletal lower limb injury in three months prior to testing.
  * Goalkeepers were excluded from the analysis

Ages: 15 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Power | 6 weeks
  Vertical jump tests are among the most common means of evaluating physical fitness in various populations. Though principally used to evaluate leg power in sports, such as basketball and football. vertical jump tests have also been used to evaluate non-athletic populations (including children (Acero et al., 2011) and elderly people (Pereira et al., 2012)), particularly because vertical jump training has been reported to improve bone mineral density (Allison, Folland, Rennie, Summers, & Brooke-Wavell, 2013). Vertical jump tests have been proposed as important for talent identification purposes, with young elite athletes displaying higher values than their non-elite counterparts.(13)
Agility | 6 weeks
  Agility is an important characteristic of team sports athletes. There is a growing interest in the factors that influence agility performance as well as appropriate testing protocols and training strategies to assess and improve this quality. Agility tests generally offer good reliability, although this may be compromised in younger participants responding to various scenarios. A human and/or video stimulus seems the most appropriate method to discriminate between standard of playing ability. Decision-making and perceptual factors are often propositioned as discriminant factors; however, the underlying mechanisms are relatively unknown.(14)
The Functional Movement Scale (FMS) | 6 weeks
  Functional (e.g., deficits in balance and strength/power performance), neural (e.g., loss of sensory/motor neurons), muscular (e.g., atrophy of type-II muscle fibers in particular), and bone-related (e.g., osteoporosis) deteriorations. Traditionally, balance and/or lower extremity resistance training were used to mitigate these age-related deficits. However, the effects of resistance training are limited and poorly translate into improvements in balance, functional tasks, activities of daily living, and fall rates.

CONTACTS AND LOCATIONS:
Overall Officials: Aamir Gul Memon, MS, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punajb, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Petway AJ, Freitas TT, Calleja-Gonzalez J, Medina Leal D, Alcaraz PE. Training load and match-play demands in basketball based on competition level: A systematic review. PLoS One. 2020 Mar 5;15(3):e0229212. doi: 10.1371/journal.pone.0229212. eCollection 2020. PMID 32134965
- [Background] Miguel M, Oliveira R, Loureiro N, Garcia-Rubio J, Ibanez SJ. Load Measures in Training/Match Monitoring in Soccer: A Systematic Review. Int J Environ Res Public Health. 2021 Mar 8;18(5):2721. doi: 10.3390/ijerph18052721. PMID 33800275
- [Background] Silva JR, Nassis GP, Rebelo A. Strength training in soccer with a specific focus on highly trained players. Sports Med Open. 2015;1(1):17. doi: 10.1186/s40798-015-0006-z. Epub 2015 Apr 2. PMID 26284158
- [Background] Taheri E, Nikseresht A, Khoshnam E. The effect of 8 weeks of plyometric and resistance training on agility, speed and explosive power in soccer players. European Journal of Experimental Biology. 2014;4(1):383-6.
- [Background] Davies G, Riemann BL, Manske R. CURRENT CONCEPTS OF PLYOMETRIC EXERCISE. Int J Sports Phys Ther. 2015 Nov;10(6):760-86. PMID 26618058
- [Background] Moreno-Perez V, Rodas G, Penaranda-Moraga M, Lopez-Samanes A, Romero-Rodriguez D, Aagaard P, Del Coso J. Effects of Football Training and Match-Play on Hamstring Muscle Strength and Passive Hip and Ankle Range of Motion during the Competitive Season. Int J Environ Res Public Health. 2022 Mar 2;19(5):2897. doi: 10.3390/ijerph19052897. PMID 35270589
- [Background] Moreno-Perez V, Campos-Vazquez MA, Toscano J, Sotos-Martinez VJ, Lopez-Del Campo R, Resta R, Del Coso J. Influence of the Weekly and Match-play Load on Muscle Injury in Professional Football Players. Int J Sports Med. 2022 Aug;43(9):783-790. doi: 10.1055/a-1533-2110. Epub 2022 Feb 21. PMID 35189659
- [Background] Maughan PC, MacFarlane NG, Swinton PA. Quantification of training and match-play load across a season in professional youth football players. International Journal of Sports Science & Coaching. 2021;16(5):1169-77.
- [Background] Morgans R, Di Michele R, Drust B. Soccer Match Play as an Important Component of the Power-Training Stimulus in Premier League Players. Int J Sports Physiol Perform. 2018 May 1;13(5):665-667. doi: 10.1123/ijspp.2016-0412. Epub 2018 Jan 2. PMID 28422525
- [Background] Horsley IG Dr, O'Donnell V, Leeder J. The epidemiology of injuries in English professional squash; A retrospective analysis between 2004 and 2015. Phys Ther Sport. 2020 Nov;46:1-6. doi: 10.1016/j.ptsp.2020.07.009. Epub 2020 Aug 5. PMID 32823248
- [Background] MOHANTA N, KALRA S, PAWARIA S. A Comparative Study of Circuit Training and Plyometric Training on Strength, Speed and Agility in State Level Lawn Tennis Players. Journal of Clinical & Diagnostic Research. 2019;13(12)
- [Background] Prvulović N, Lilić A, Hadžović M. THE PREVALENCE OF FOOT DEFORMITIES IN ATHLETES WITH VARIOUS SPORTS BACKGROUNDS. Facta Universitatis Series: Physical Education and Sport. 2021:667-79.
- [Background] Balsalobre-Fernandez C, Glaister M, Lockey RA. The validity and reliability of an iPhone app for measuring vertical jump performance. J Sports Sci. 2015;33(15):1574-9. doi: 10.1080/02640414.2014.996184. Epub 2015 Jan 2. PMID 25555023
- [Background] Paul DJ, Gabbett TJ, Nassis GP. Agility in Team Sports: Testing, Training and Factors Affecting Performance. Sports Med. 2016 Mar;46(3):421-42. doi: 10.1007/s40279-015-0428-2. PMID 26670456
- [Background] Granacher U, Gollhofer A, Hortobagyi T, Kressig RW, Muehlbauer T. The importance of trunk muscle strength for balance, functional performance, and fall prevention in seniors: a systematic review. Sports Med. 2013 Jul;43(7):627-41. doi: 10.1007/s40279-013-0041-1. PMID 23568373